CLINICAL TRIAL: NCT00018785
Title: Living-Related Donor Bone Marrow Immunoregulation in Kidney Transplants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMMU-035-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Kidney Disease
Keywords: kidney transplantation; immunosuppression; bone marrow
MeSH Terms: conditions — Kidney Diseases

INTERVENTIONS:
Procedure: donor bone marrow infusion

SUMMARY:
Diabetes and end-stage kidney, liver and heart disease are prominent health issues among veteran patients. Successful solid organ transplantation in the absence of chronic immunosuppressive therapy (specific acquired immunological tolerance) is a desirable therapeutic option. This project extends recent observations supporting the use of concommitant donor bone marrow cell infusion as a means of modulating the immune response in kidney transplantation, thereby allowing a substantial decrease or withdrawal of potentially toxic immunosuppressive drugs.

ELIGIBILITY:
Living related donor kidney transplant recipients and the living related donors.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-10; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Ricordi, M.D.; Andreas Tzakis, M.D.; Violet Esquenazi, Ph.D.; Keith Zucker, Ph.D.
Locations (1):
- VAMC Miami, Miami, Florida, United States